CLINICAL TRIAL: NCT05601479
Title: Preventive Effect of Acetyl-L-carnitine on Oxaliplatin-induced Peripheral Neuropathy： A Randomized, Controlled, Open-label, Phase 2 Trail
Brief Title: Preventive Effect of Acetyl-L-carnitine on Oxaliplatin-induced Peripheral Neuropathy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, Wang Chunlin, Clinical Associate professor, Nanfang Hospital, Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NFEC-2022-362
Record Dates: First submitted 2022-10-25; First posted 2022-11-01 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Acetylcarnitine; Chemotherapy-induced Peripheral Neuropathy
MeSH Terms: interventions — Acetylcarnitine

STUDY DESIGN:
Masking Description: This study was an open-label, unblinded study. Both participants were aware of their enrollment status.Scale evaluators, nerve conduction velocity measurement testers during the study did not know the grouping of subjects. The collected data were submitted to statistical experts who were unaware of the group assignments for statistical analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acetyl-L-carnitine group(ALC group) (Experimental): At the beginning of the first chemotherapy of the oxaliplatin regimen, acetyl-L-carnitine 500mg will be given orally three times daily for 24 weeks.
  Interventions: Drug: Acetyl-L-carnitine
- Blank Control group (No Intervention): No drugs for the prevention and treatment of peripheral neuropathy will be given.

INTERVENTIONS:
Drug: Acetyl-L-carnitine — At the beginning of the first chemotherapy of the oxaliplatin regimen, Acetyl-L-carnitine 500mg will be given orally three times daily for 24 weeks. If subjects discontinue oxaliplatin-containing chemotherapy for various reasons (e.g., allergy to oxaliplatin), they will continue taking acetyl-L-carnitine until 24 weeks (unless acetyl-L-carnitine intolerance or other conditions interfere with medication).
  Other Names: Chinese Food and Drug Administration H20180021
  Arms: Acetyl-L-carnitine group(ALC group)

SUMMARY:
With the prolongation of the overall survival time of patients with malignant tumors, the influence of oxaliplatin on the quality of life of patients with malignant tumors has gradually become prominent. Studies have shown that acetyl-L-carnitine can improve the energy metabolism of neurotransmitters and inhibit the release of glutamine in the intersynaptic space to reduce pain. Large-scale clinical studies have approved it as a treatment for diabetic peripheral neuropathy. Some small model studies have also found that acetyl-L-carnitine has a definite therapeutic effect on peripheral neurological lesions induced by chemotherapy. The aim of this study is to investigate the safety and efficacy of acetyl-L-carnitine in the prevention of oxaliplatin-induced peripheral neuropathy. The study was divided into an experimental group and a control group. The experimental group was given acetyl-L-carnitine orally, and the researchers regularly evaluated the symptoms and electrophysiological indicators related to peripheral neuropathy. If there is a severe adverse reaction related to acetyl-L-carnitine, the drug should be discontinued and the symptomatic treatment should be given. After the completion of the study, the statistical calculation and analysis will be used to estimate whether the preventive and therapeutic effect of acetyl-L-carnitine on oxaliplatin-induced peripheral neuropathy was statistically significant.

DETAILED DESCRIPTION:
1. Background 1.1 Epidemiological overview of oxaliplatin-induced peripheral neuropathy Gastrointestinal cancer is the most common malignant tumor in the world, mainly including Gastric cancer (GC), Colorectal cancer (CRC) and so on. In the past decade, with the development of diagnosis and treatment technology, the survival time of patients with gastrointestinal malignant tumors has significantly increased, among which platinum-based chemotherapy drugs play an important role. Oxaliplatin (OXA) is the third generation of platinum-based chemotherapy drugs, which is characterized by high efficiency, low toxicity and broad spectrum, and has become the main drug in the treatment of a variety of gastrointestinal malignant tumors. However, with the widespread application of oxaliplatin, its related adverse reactions have gradually become prominent. Oxaliplatin induced peripheral neuropathy (OIPN) is a dose-limiting adverse reaction, which can be usually divided into acute and chronic OIPN according to the severity of onset. Acute OIPN mainly manifests as paresthesia, such as tingling and numbness induced or aggravated by cold stimulation, which usually appears several hours after administration and disappears within a few days. Chronic OIPN is associated with dose accumulation and develops in approximately 70% of patients receiving OXA . After the cumulative OXA dose of 540-850 mg/m2, equivalent to 9-10 cycles of 85 mg/m2 or 6 cycles of 130 mg/m2, most patients had peripheral neuropathy symptoms that did not relieve between treatment intervals. In addition to tingling and numbness similar to acute OIPN, symptoms such as hypoesthesia of proprioception and/or fine touch and ataxia that seriously affect the quality of daily life can also occur.

   1.2 Treatment status of oxaliplatin-induced peripheral neuropathy at home and abroad At present, the specific mechanism of OIPN is still inconclusive. Over the years, researchers have proposed a variety of possible mechanisms around Dorsal root ganglion (DRG), including: abnormal opening and closing of ion channels, activation and inactivation of transporters, nuclear dysfunction, abnormal mitochondrial DNA function, and axonal degeneration. A variety of drug studies for the prevention and treatment of OIPN have been carried out based on the above mechanisms. Only Duloxetine is recommended by the American Society of Clinical Oncology (ASCO) for moderate prevention of OIPN at present, because it often fails to achieve ideal preventive effect in clinical application due to drug side effects and efficacy.Therefore, drug withdrawal is the main option to limit the progression of OIPN when severe neuropathy occurs. According to ASCO's updated guidelines for the prevention and treatment of chemotherapy-induced peripheral neuropathy, calcium-magnesium mixture, calmangafodipir, L-carnosine , alpha-lipoic acid, ganglioside (GM-1), metformin, venlafaxine, pregabalin, vitamin E/B, minocycline and other drugs have been tried to prevent CIPN caused by oxaliplatin, but they are all in clinical trials at various stage, and none of them has been proven effective. In addition to drug therapy, there are many studies using a variety of physical therapies, such as acupuncture, cryotherapy, compression therapy, exercise therapy, etc. Traditional Chinese medicine (TCM) has adopted its unique treatment methods, such as classical prescription, self-made prescription, traditional Chinese medicine injection, acupuncture, fumigation and acupoint application, but the preventive efficacy remains unclear.

   1.3 Theoretical basis for the prevention of oxaliplatin-induced peripheral neuropathy by acetyl-L-carnitine Acetyl-L-carnitine is the acetylation product of L-carnitine, which can penetrate the blood-brain barrier and decompose into acetyl group and L-carnitine after entering the central nervous system. L-carnitine plays a role in transporting long-chain fatty acids between the inner and outer membranes of mitochondria, participating in fatty acid β-oxidation and providing energy for cells. Acetyl groups are directly involved in the synthesis of acetyl coenzyme A(acetyl-CoA) and other important metabolic mediators and indirectly in the tricarboxylic acid cycle. In addition, studies have shown that acetyl groups can also act on mGlu2 receptors located in the presynaptic membrane of the posterior horn of the spinal cord to alleviate pain by reducing the release of the excitatory amino acid transmitter glutamate. L-carnitine and acetyl groups are both physiological components of the human body, so acetyl-L-carnitine has no obvious toxic and side effects. Clinical trials of acetyl-L-carnitine in China occasionally reported mild excitement, but the symptom could be eliminated by reducing the dose. The total incidence of adverse reactions was 6.84% (8/117), mainly manifested as gastrointestinal symptoms (belching, nausea, abdominal distension, dizziness, abnormal liver function, weight loss, etc.), most of them were mild (7 cases), and 1 case was moderate. There were no sequelae after remission.

   At present, the approved indication of acetyl-L-carnitine in China is diabetic peripheral neuropathy. Acetyl-L-carnitine has also been used in the treatment of chemotherapy-induced peripheral neuropathy (CIPN) in small clinical studies, and the results suggest that it has good preventive effect. However, the subjects of this study were diverse, the design was not a single chemotherapy drug, and the inclusion criteria were patients who had developed peripheral neuropathy. Therefore, our study intends to simplify the study object to OIPN caused by oxaliplatin and use it in the prevention stage in order to avoid OIPN.

   In summary, acetyl-L-carnitine has a mature clinical application, high safety, and low price. Some studies have suggested that it has a therapeutic effect on chemotherapy-induced peripheral neuropathy, and is worthy of further clinical research as a potential drug for the prevention of OIPN induced by oxaliplatin.
2. Research Purpose 2.1 Main Research Purpose To evaluate the efficacy of acetyl-L-carnitine in the prevention of oxaliplatin-induced chronic peripheral neuropathy (OIPN).

   2.2 Secondary Research Purpose To evaluate the safety of acetyl-L-carnitine in the prevention of oxaliplatin-induced chronic peripheral neuropathy (OIPN).
3. Study end point 3.1 Primary end point To evaluate the preventive effect of acetyl-L-carnitine on OIPN in patients with gastrointestinal cancer after receiving oxaliplatin-based chemotherapy, and compare the incidence of OIPN in the two groups (acetyl-L-carnitine group and blank control group) after 6 months of oxaliplatin-based chemotherapy. Because there is no uniform diagnostic criteria for all chemotherapy-induced peripheral neuropathy including OIPN, different questionnaires are used to grade the severity in the world. In order to ensure the accuracy and consistency of the diagnosis of OIPN in this study, the following diagnostic criteria were used in combination with similar research standards:1)The expected numbness, pain and other symptoms occurred after receiving oxaliplatin treatment. 2)A score of 3 or higher on section A (medical history) and 2 or higher on section B (physical examination) on the Michigan Neuropathy Assessment Scale. 3)Exclusion of other causes of peripheral neuropathy (In this study, subjects will be screened for exclusion of other causes of peripheral neuropathy before enrollment).

3.2 Secondary study end Point

1)To compare the severity of OIPN (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Chemotherapy-Induced Peripheral Neuropathy 20-Item Scale[EORTC QLQ-CIPN20], nerve conduction velocity measurement including compound muscle action potentials [CMAP] and compound muscle action potentials[SNAP] ) between the acetyl-L-carnitine group and the blank control group after 6 months of oxaliplatin-based chemotherapy.2)The occurrence time of OIPN was compared between the two groups.3)Comparison of the effects of acetyl-L-carnitine on tumor prognosis (progression-free survival and overall survival) between the two groups.

4.Experimental design This study is a randomized, controlled and open-label phase 2 clinical study.

1. Appropriate subjects will be selected according to the inclusion and exclusion criteria. Subjects who met the inclusion and exclusion criteria will be randomly divided into the acetyl-L-carnitine test group and the blank control group at a ratio of 1:1 by envelope drawing method until 100 subjects were included. At the beginning of the first chemotherapy of oxaliplatin regimen, acetyl-L-carnitine 500mg will be given orally three times daily for 24 weeks. If subjects discontinue oxaliplatin-containing chemotherapy for various reasons (e.g., allergy to oxaliplatin), they will continue taking acetyl-L-carnitine until 24 weeks (unless acetyl-L-carnitine intolerance or other conditions interfere with medication).
2. Subjects will be treated with oxaliplatin-containing regimens (mFOLFOX6, CapeOX, FOLFOXIRI, and so on) according to clinical practice.
3. QLQ-CIPN20 sensory scale and nerve conduction study (NCV) will be used to evaluate the peripheral nerve status at baseline, 12, 24 and 48 weeks after enrollment.
4. Participants could withdraw from the trial if they were deemed by the investigator to be unfit to continue the trial, such as intolerable toxicity, loss to follow-up, withdrawal of consent and refusal to provide further information.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* The Eastern Cooperative Oncology Group (ECOG) performance status was 0 or 1
* The predicted survival time was ≥12 months
* Subjects will receive oxaliplatin-containing regimens, including
* mFOLFOX6 scheme Oxaliplatin: 85mg/m2 was infused intravenously for 2 hours, day 1; Leucovorin calcium: 400 mg/m2 was infused intravenously for 2 hours, 1 day; 5 - Fluorouracil: After 400mg/m2 intravenous bolus on day 1, then 1200mg (m2•d) continuous intravenous pump infusion (total 2400mg/m2, infusion 46-48h); Chemotherapy will be performed every 2 weeks for 12 cycles.
* CapeOX scheme Oxaliplatin: 130 mg/m2 was infused intravenously for 2 hours, day 1; capecitabine: 1000 mg/m2 orally, bid, 1-14 days; Chemotherapy will be performed every 3 weeks for 8 cycles.
* FOLFOXIRI scheme Irinotecan: 165 mg/m2 was infused intravenously, day 1; Oxaliplatin:85mg/m2 was infused intravenously, day 1; Leucovorin calcium: 400 mg/m2 was infused intravenously, day 1; 5 - Fluorouracil: The total dose of 5-FU was 2400-3200 mg/m2, and the intravenous infusion lasted for 48 hours, day 1; Chemotherapy will be performed every 2 weeks for 12 cycles.
* Laboratory values within 7 days before enrollment should meet the following criteria:

Blood routine: neutrophil count (ANC) ≥1.5×109/L, platelet count (PLT) ≥100×109/L, hemoglobin (HGB) ≥80g/L; Liver function: serum total bilirubin (TBIL) ≤ 1.5 times upper limit of normal (ULN), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 times upper limit of normal; Renal function: creatinine clearance (CCr) ≥ 50ml/min;

* Patients should voluntarily participant in the study, provide written informed consent, and adhere to protocol-specified visits and procedures.

Exclusion Criteria:

* Participating in other interventional clinical studies (unless participating in an observational study or in the follow-up phase of an interventional study);
* Hyponatremia, hypokalemia, hyperchloremic acidosis, adrenal failure and adrenocortical insufficiency (Addison's disease), hepatic coma, diabetes mellitus, brain or leptomeningeal metastases;
* Patients who has previously received neurotoxic chemotherapy such as taxanes, vinca alkaloids, or cisplatin and received any other medication specifically for the treatment or prevention of neuropathy;
* Patients with peripheral neuropathy (confirmed by nerve conduction velocity measurements) due to other causes (such as radiation or malignant plexopathy, lumbar or cervical radiculopathy, vitamin B12 deficiency, or diabetes) before chemotherapy;
* History of alcohol dependence or concomitant use of other drugs known to affect serotonin levels;
* Having cardiovascular clinical symptoms or disease that is not well controlled;
* The presence of a mental illness or substance abuse condition that may have affected adherence to trial requirements;
* Women who are pregnant or lactating;
* There are medical history, disease, treatment, or laboratory abnormalities that may interfere with the results of the trial, prevent the participant from participating in the study throughout, or the researcher believes that participation in the study is not in the best interests of the participant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of OIPN | week 24 after enrollment
  To evaluate the preventive effect of acetyl-L-carnitine on OIPN in patients with gastrointestinal 24 weeks of oxaliplatin-based chemotherapy.

SECONDARY OUTCOMES:
Severity of OIPN | week 24 after enrollment
  The severity of OIPN was compared between the acetyl-L-carnitine group and the blank control group after 24 weeks of oxaliplatin-based chemotherapy.
Time of occurrence | week12, week 24, week 48 after enrollment
  Comparison the occurrence time of OIPN between the two groups.
The prognosis of tumor | week12, week 24, week 48 after enrollment
  To explore the effect of acetyl-L-carnitine on the prognosis of patients with tumor.

CONTACTS AND LOCATIONS:
Overall Officials: Chunlin Wang, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital, Southern Medical University/The First School of Clinical Medicine, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Campone M, Berton-Rigaud D, Joly-Lobbedez F, Baurain JF, Rolland F, Stenzl A, Fabbro M, van Dijk M, Pinkert J, Schmelter T, de Bont N, Pautier P. A double-blind, randomized phase II study to evaluate the safety and efficacy of acetyl-L-carnitine in the prevention of sagopilone-induced peripheral neuropathy. Oncologist. 2013;18(11):1190-1. doi: 10.1634/theoncologist.2013-0061. Epub 2013 Oct 8. PMID 24105751
- [Result] Hershman DL, Unger JM, Crew KD, Minasian LM, Awad D, Moinpour CM, Hansen L, Lew DL, Greenlee H, Fehrenbacher L, Wade JL 3rd, Wong SF, Hortobagyi GN, Meyskens FL, Albain KS. Randomized double-blind placebo-controlled trial of acetyl-L-carnitine for the prevention of taxane-induced neuropathy in women undergoing adjuvant breast cancer therapy. J Clin Oncol. 2013 Jul 10;31(20):2627-33. doi: 10.1200/JCO.2012.44.8738. Epub 2013 Jun 3. PMID 23733756
- [Result] Sun Y, Shu Y, Liu B, Liu P, Wu C, Zheng R, Zhang X, Zhuang Z, Deng Y, Zheng L, Xu Q, Jiang B, Ouyang X, Gao J, Xu N, Li X, Jiang S, Liang C, Yao Y. A prospective study to evaluate the efficacy and safety of oral acetyl-L-carnitine for the treatment of chemotherapy-induced peripheral neuropathy. Exp Ther Med. 2016 Dec;12(6):4017-4024. doi: 10.3892/etm.2016.3871. Epub 2016 Nov 4. PMID 28105133
- See also: EORTC QLQ-CIPN20 — http://www.eortc.org/app/uploads/sites/2/2018/08/Specimen-CIPN20-English.pdf
- See also: Common Terminology Criteria for Adverse Events, CTCAE, version 5.0 — http://ctep.cancer.gov/protocolDevelopment/electronic_applications/ctc.htm